CLINICAL TRIAL: NCT04722198
Title: Effects of Lactobacillus Plantarum PS128 on Symptoms of Early-onset Parkinson's Disease: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Lu Neurological Clinic (Other)
Responsible Party: Principal Investigator, CHIN-SONG LU, Professor, Professor Lu Neurological Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PS128-04
Record Dates: First submitted 2021-01-15; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Early Onset Parkinson Disease
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PS128 (Experimental): Each PS128 capsule contained >1 × 10^10 colony forming units (CFU) with microcrystalline cellulose and weights 425 ± 25 mg
  Interventions: Dietary Supplement: PS128

INTERVENTIONS:
Dietary Supplement: PS128 — daily ingestion 2 capsules of Lactobacillus plantarum PS128 (>10 billion CFU/capsule)

SUMMARY:
This study is designed to examine L. plantarum PS128 can improve symptoms in early onset PD patients. L. plantarum PS128 is a psychobiotic that regulates the level of dopamine in specific brain regions. Patients with early onset PD will receive PS128 treatment for 12 weeks. Symptoms of PD will be clinically evaluated before and after the treatment, and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Early Onset Parkinson's Disease, EOPD
* at least 9 years education
* age between 20 and 80 years old

Exclusion Criteria:

* Patients on antibiotics within the preceding one month
* Patients using of other probiotic products (sachet, capsule or tablet) within the preceding two weeks
* Have undergone surgery of liver, bladder, or gastrointestinal tract
* Have current or history of inflammatory bowel disease
* Have history of cancer
* Known allergy to probiotics
* Patients with comorbid dementia (Mini-Mental State Examination score ≤ 26) or major depression (The Beck Depression Inventory-II score ≥ 29)
* Have received deep brain stimulation
* Patients receiving artificial enteral or intravenous nutrition
* Diagnosed before 40 years old
* Poor control of other chronic diseases
* Not eligible judged by PI

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
UPDRS III | 12 weeks
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients.
  The PART III is Motor sections.
MHY | 12 weeks
  The Hoehn and Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress.
  The modified Hoehn and Yahr scale included stages 1 through 5. to help describe the intermediate course of the disease.
TUG | 12 weeks
  Observe the patient's postural stability, gait, stride length, sway and test cut-off times.

SECONDARY OUTCOMES:
UPDRS I-IV | Baseline and Post-12 weeks
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients.
  The UPDRS scale consists of the following five segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, 4) Modified Hoehn and Yahr Scale, and 5) Schwab and England ADL scale.
SCL-90-R | Baseline and Post-12 weeks
  The Symptom Checklist-90-Revised instrument helps evaluate a broad range of psychological problems and symptoms of psychopathology.
  The SCL-90-R is normed on individuals 13 years and older. It consists of 90 items and takes 12-15 minutes to administer.
CPSQI | Baseline and Post-12 weeks
  The Chinese Version of the Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.The maximum total score is 21. A higher score reflects more poor sleep quality.
VAS-GI | Baseline and Post-12 weeks
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
PGIC | Post-12 weeks
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Lu Neurological Clinic, Taoyuan, Guishan Dist., Taiwan